CLINICAL TRIAL: NCT05439889
Title: Follow-up Study on Chronic Myeloid Leukemia Patients Achieving Treatment-free Remission
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202202074RINB
Record Dates: First submitted 2022-06-15; First posted 2022-06-30 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Chronic Myeloid Leukemia, BCR/ABL-Positive
Keywords: Chronic myeloid leukemia; Treatment free remission
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent years, the goal of stopping drug therapy, also known as treatment-free remission (TFR), is emerging as one of the management goals of chronic myeloid leukemia (CML) therapy. Because there is no available data on Asian patients with CML undergoing tyrosine kinase inhibitor discontinuation (TKI), the investigators plan to recruit chronic phase CML patients with deep treatment response and good medical compliance in Taiwan to evaluate the feasibility, safety and clinical consequences of TKI discontinuation.

DETAILED DESCRIPTION:
1. Primary goal: To evaluate the feasibility, safety and clinical consequences of TKI discontinuation in chronic phase CML(CP-CML) patients with deep treatment response and good medical compliance in Taiwan

2. Molecular response monitoring:

1. After discontinuation of TKI therapy, participants will receive monthly molecular monitoring of BCR-ABL transcript levels by real-time quantitative polymerase chain reaction (RT-qPCR) for one year, every two months for the second year and every three months thereafter.
2. If loss of major molecular response (MMR) (BCR-ABL transcript level ⩽ 0.1% IS) is detected at any time point post TKI discontinuation, the participant should receive repeated testing within two weeks. If loss of MMR is confirmed, TKI should be resumed within four weeks
3. RT-qPCR of BCR-ABL would be ordered every four weeks until MR4 (BCR-ABL transcript level ⩽ 0.01% IS) is re-established, and then every 12 weeks indefinitely.
4. For patients who fails to achieve MMR again within three months after TKI is re-initiated, BCR-ABL kinase domain mutation testing would be performed

ELIGIBILITY:
Inclusion Criteria:

1. The participant should be an adult (age ⩾20 years) with CP-CML.
2. The BCR-ABL fusion should be in the form of either e13a2 or e14a2 (p210)
3. The participant should not have documented resistance to a 2nd-generation TKI (Nilotinib or Dasatinib)
4. The participant should have received ≥ 5 years of consecutive treatment with imatinib, or ≥ 4 years of consecutive treatment with a 2nd-generation TKI (Nilotinib or Dasatinib)
5. The participant should have achieved MR4.5 (BCR-ABL ⩽0.0032% IS) or undetectable disease in the peripheral blood or bone marrow, for ≥ 2 years, which is documented on ≥ 4 separate tests performed ≥ 3 months apart.
6. Access to a reliable qPCR-based BCR-ABL test with a sensitivity of detecting of at least MR4.5.

Exclusion Criteria:

1. After evaluation, the participant is deemed to be ineligible by the investigator of this study.
2. The participant has no intention to be recruited into this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with CP-CML and are regularly followed up at National Taiwan University Hospital (NTUH) or at the branch hospitals of the NTUH healthcare system
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2028-08-11 (Estimated); Study Completion 2032-08-11 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who were in major molecular response (MMR) without re-initiation of treatment | at week 48 of tyrosine kinase inhibitor (TKI) discontinuation
  Real-time quantitative polymerase chain reaction (RT-qPCR) would be done to determined the transcript level of BCR-ABL fusion gene in peripheral blood samples

SECONDARY OUTCOMES:
The proportion of patients who were in MR4.5 (BCR-ABL transcript level ⩽0.0032% IS) and off treatment | at week 48 of TKI discontinuation
  Real-time quantitative polymerase chain reaction (RT-qPCR) would be done to determined the transcript level of BCR-ABL fusion gene in peripheral blood samples
Treatment-free survival | From the start of TKI discontinuation until the earliest occurrence of any of the following: loss of MMR, restart of TKI for any reason, progression to accelerated phase/blast phase, or death of any cause, assessed up to 60 months
The proportion of patients who reachieved of MMR after TKI restart | qPCR of BCR-ABL would be checked every four weeks until MR4 is re-established, and then every 12 weeks until study completion (week 240).
  Real-time quantitative polymerase chain reaction (RT-qPCR) would be done to determined the transcript level of BCR-ABL fusion gene in peripheral blood samples
The proportion of patients who reachieved of MR4.5 after TKI restart | qPCR of BCR-ABL would be checked every four weeks until MR4 is re-established, and then every 12 weeks until study completion (week 240).
  Real-time quantitative polymerase chain reaction (RT-qPCR) would be done to determined the transcript level of BCR-ABL fusion gene in peripheral blood samples
Incidence and severity of treatment-related adverse events [Safety and Tolerability] | Evaluation of AEs would be conducted on an ongoing basis on study until 30 days after the last day of TFR
  Adverse events (AEs) would be assessed according to the CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan